CLINICAL TRIAL: NCT04779853
Title: Seroprevalence of Pertussis Among Healthy Children and Adolescents in Kazakhstan: A Cross-Sectional Study
Brief Title: Seroprevalence of Pertussis Among Healthy Children and Adolescents in Kazakhstan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scientific and practical center of sanitary and epidemiological expertise and monitoring (Other)
Responsible Party: Sponsor
Other Study IDs: PER00075
Record Dates: First submitted 2021-01-25; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Pertussis
Keywords: pertussis; seroprevalence; immunity; antibodies; Kazakhstan; vaccination
MeSH Terms: conditions — Whooping Cough | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — This study will be a cross-sectional serosurvey of anti-PT levels in a sample of the population. The study will be conducted in the cities of Aktobe, Karaganda, Taldykorgan, and Shymkent. Enrollment will be done in health centers and pediatric hospitals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pertussis antibodies testing will be conducted at the Reference Laboratory in NPCCEEM: serum samples will be taken and tested by enzyme-linked immunoassay (ELISA) using the SAVYON SeroPertussisTM kits (Savyon Diagnostics Ltd, Israel).
  Interventions: Diagnostic Test: Blood samples for pertussis antibody testing

INTERVENTIONS:
Diagnostic Test: Blood samples for pertussis antibody testing — Blood samples will be sent to the laboratories of the National Centers of Expertise within 24-48 hours of blood collection. The samples will be transferred to the reference laboratory of SPCSEEM in Almaty, Kazakhstan. Serum samples will be stored in the reference laboratory at a temperature of -20 C.

SUMMARY:
Seroprevalence of pertussis among older children and adolescents in Kazakhstan: A cross sectional study.

Justification: to describe the distribution of anti-pertussis toxin (PT) antibodies (IgA and IgG) in a population aged 10-18 years old according to sociodemographic characteristics, vaccination history, and risk factors of pertussis infection.

DETAILED DESCRIPTION:
Pertussis due to infection with Bordetella pertussis (B pertussis) is a well-known cause of persistent cough primarily affecting infants and young children. Repeated administration of the vaccine is often needed to reduce the disease burden and control its transmission. At this time, no data are available on the epidemiology of pertussis in adolescents and adults in Kazakhstan.

The aim of the present study is to estimate the prevalence of pertussis infection in different age groups in Kazakh children and adolescents using the anti-pertussis toxin (PT) antibodies (IgA and IgG) as specific marker of pertussis infection or vaccination. The serosurvey will be conducted in 4 different regions: Aktobe, Karaganda, Taldykorgan, and Shymkent.

Participants (≥ 10 years & < 19 years) attending the study centers will be asked to participate in the study. The adolescent participants and the parents/guardian(s) of all participants will be informed about the procedures and data handling. Written informed consent from one parent/guardian needs to be obtained by the physician before any blood samples can be taken.

Upon obtaining informed consent for participant parent/guardian, the study coordinator will complete an investigation form (IF) for each participant and collect serum samples. The specimens will be coded by a unique participant number and delivered to the laboratory in charge of the assay. The specimens will be used for serological analyses.

ELIGIBILITY:
Inclusion Criteria:

10-18 years old

* Informed consent obtained from parents or guardian(s) and assent from patient.
* Enrollment following a visit at the study center.
* Documented vaccination history

Exclusion Criteria:

Inclusion criteria:

* 10-18 years old
* Informed consent obtained from parents or guardian(s) and assent from patient.
* Enrollment following a visit at the study center.
* Documented vaccination history

Exclusion criteria:

* ≤10 years and ≥ 19 years
* Pertussis immunization during the last 12 months
* No informed consent obtained from one parent or guardian.
* Immunocompromised patients
* Patients with acute infectious diseases

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants (≥ 10 years & < 19 years) attending the study centers will be asked to participate in the study. The adolescent participants and the parents/guardian(s) of all participants will be informed about the procedures and data handling. Written informed consent from one parent/guardian needs to be obtained by the physician before any blood samples can be taken.
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-10-17 (Estimated); Study Completion 2022-07-05 (Estimated)

PRIMARY OUTCOMES:
The anti-PT IgG and Ig A concentrations (in IU/ml) in the population sample. | 25.01.2021-17.10.2021
  To estimate the prevalence of recent infection Bp infection, using increased anti-PT antibody levels as markers of Bp infection in the serology test.

SECONDARY OUTCOMES:
The prevalence of recent Bp infection in the test in the selected population sample stratified by demographic and socio-economic criteria, vaccination history, and risk of infection. | 25.01.2021-17.10.2021
  To evaluate the risk factors associated with higher seroprevalence of pertussis.

OTHER OUTCOMES:
• Adherence to vaccination status defined as the. number and timeliness of doses received and potential exposure to booster vaccination as well as the concordance with the Kazakh vaccination status. | 25.01.2021-17.10.2021
  • To evaluate the compliance with recommended vaccination schedule in study participants

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific and Practical Center of Sanitary and Epidemiological Expertise and Monitoring, Almaty, Kazakhstan

DOCUMENTS (4):
  • Study Protocol (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT04779853/Prot_000.pdf
  • Informed Consent Form (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT04779853/ICF_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT04779853/SAP_002.pdf
  • Statistical Analysis Plan: Survey (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT04779853/SAP_003.pdf